CLINICAL TRIAL: NCT06584422
Title: Community-Embedded, Layperson-Supported Digital Mental Health Intervention for Homebound Older Adults With Depression: A Type 1 Hybrid Effectiveness- Implementation RCT
Brief Title: Empower@Home: Hybrid Effectiveness-Implementation Randomized Controlled Trial (RCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); NYU Silver School of Social Work (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Xiaoling Xiang, PhD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00254688; R01MH137064 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Depression
Keywords: Cognitive behavioral therapy; Older Adults; Internet-based intervention; Depression; Social isolation
MeSH Terms: conditions — Depression; Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding interventionalists and participants is not possible, given the nature of the intervention. However, assessment staff will be blinded when possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empower@Home supported by aging service providers (Experimental): Participants will be provided with access to a 9-session online program called Empower@Home, a self-help intervention based on cognitive behavioral therapy principles. The intervention has three components: 9 interactive self-paced online sessions, printed workbook that goes along the online sessions for exercises and homework, and telephone coaching by a trained staff from a social service agency serving older adults. Participants will have up to 12 weeks to try to complete the program with the support of a trained coach.
  Interventions: Behavioral: Empower@Home: An online cognitive-behavioral therapy self-care program for geriatric depression
- Attention call with friendly visitors (Other): Participants will receive enhanced care as usual, including care as usual from their social service provider and a psycho-educational handout. In addition, they will receive telephone friendly calls from a research staff every other week to mimic the human interactions provided by coaches in the experimental group.
  Interventions: Other: Telephone friendly visits

INTERVENTIONS:
Behavioral: Empower@Home: An online cognitive-behavioral therapy self-care program for geriatric depression — Empower@Home is an online self-help intervention based on cognitive behavioral therapy principles designed to treat depressive symptoms in older adults. The intervention has three components: 9 interactive self-paced online sessions, printed workbook that goes along the online sessions for exercises and homework, and telephone coaching by a trained staff from a social service agency serving older adults. The online sessions contain entertainment elements in the form of a character-driven story of a homebound older adults, video-based psycho-educational content, voice-over instructions, interactive exercises, and weekly home practice assignments.
  Arms: Empower@Home supported by aging service providers
Other: Telephone friendly visits — Participants in the waitlist control group will receive attention control through biweekly telephone-friendly visitors. Trained project staff will call participants to provide companionship, emotional support, and a friendly conversation. In addition, the callers will conduct a biweekly assessment of depressive symptoms using the patient health questionnaire (PHQ-9), to mirror the biweekly in-app PHQ-9 assessments with the experimental group.
  Arms: Attention call with friendly visitors

SUMMARY:
This study is a randomized Type I hybrid effectiveness-implementation trial aimed at evaluating the effectiveness of Empower@Home, an internet-delivered cognitive-behavioral therapy (CBT) program supported by aging service providers, in comparison to enhanced usual care for homebound older adults with depressive symptoms. A total of 256 participants will be randomly assigned to either the treatment group (Empower@Home) or the control group (enhanced usual care) in a 1:1 allocation ratio, with randomization stratified by participating agencies.

The primary aim of this study is to determine the clinical effectiveness of the Empower@Home program. It is hypothesized that participants receiving Empower@Home will show greater improvements in depressive symptoms at 12, 24, and 36 weeks after entering the study compared to those receiving enhanced usual care. Additionally, treatment moderators will be explored and a cost-effectiveness analysis will be conducted to assess the economic viability of the intervention.

The second aim is to investigate the mechanisms of change facilitated by the intervention using a mixed-methods approach. Causal mediation analysis will examine whether the acquisition of CBT skills, reduction in cognitive distortions, and increased behavioral activation, as well as participant engagement and the therapeutic alliance with the coach, mediate the treatment effects. Qualitative interviews with participants will be conducted to provide deeper insights into these mechanisms and enhance the interpretation of the mediation analysis.

The third aim focuses on evaluating the implementation process using the updated Consolidated Framework for Implementation Research (CFIR). This will involve a qualitative process evaluation to identify barriers and facilitators to the implementation of Empower@Home, drawing on perspectives from multiple stakeholders.

DETAILED DESCRIPTION:
This study is a randomized Type I hybrid effectiveness-implementation trial designed to evaluate the clinical effectiveness and implementation process of Empower@Home, an internet-delivered cognitive-behavioral therapy (CBT) program tailored for homebound older adults with depressive symptoms. The trial compares Empower@Home, supported by aging service providers, to an enhanced usual care condition. The study involves 256 participants who will be randomly assigned to either the treatment or control group, with randomization stratified by agency.

Rationale: Depression is a significant public health concern among homebound older adults, with approximately 50% experiencing clinically significant depressive symptoms and 14% facing major depression-rates significantly higher than those of non-homebound counterparts. Homebound older adults often encounter barriers to accessing traditional mental health services, including physical disabilities, socioeconomic disadvantages, and racial or ethnic minority status. Empower@Home addresses these challenges by leveraging the existing workforce of aging service providers to support digital mental health interventions (DMHIs).

Intervention: Empower@Home is a nine-session, computerized CBT program enhanced with entertainment elements to increase engagement. The program is specifically designed for homebound older adults, incorporating age-relevant examples and a simplified user interface. It includes features such as a character-driven storyline, short videos, and interactive exercises to facilitate learning and engagement. The program is supported by lay coaches-aging service providers trained to offer weekly support calls, enhancing program adherence and personalization.

Study Aims:

Effectiveness: The primary aim is to determine the clinical effectiveness of Empower@Home compared to enhanced usual care. The hypothesis is that participants in the Empower@Home group will show greater improvements in depressive symptoms at 12, 24, and 36 weeks post-enrollment. Secondary clinical outcomes include improvements in anxiety, loneliness, social support, quality of life, disability burden, and pain severity.

Mechanisms of Change: The study will also explore the mechanisms through which the intervention produces change. Using a mixed-methods approach, the study will investigate whether CBT-related factors (e.g., skill acquisition, behavioral activation), engagement-related factors (e.g., narrative engagement), and coach-related factors (e.g., therapeutic alliance) mediate treatment effects. Qualitative interviews will complement these findings by providing participant perspectives on how the program facilitated behavioral change.

Implementation: The study will assess the implementation process using the updated Consolidated Framework for Implementation Research (CFIR). This qualitative process evaluation will identify barriers and facilitators to implementation from the perspectives of multiple stakeholders, including older adults, coaches, and agency staff. Data will be collected through interviews, meeting minutes, field observations, and other relevant sources, and analyzed using both traditional qualitative methods and natural language processing techniques.

Study Design: Participants will be recruited from 3 to 4 aging service agencies that serve as implementation sites. These agencies represent diverse service delivery models, enhancing the study's external validity. Participants will undergo remote assessments via phone at baseline, post-intervention, and follow-up intervals at 12, 24, and 36 weeks. The study will also employ a cost-effectiveness analysis, evaluating the economic viability of the Empower@Home program from a public healthcare payer perspective.

Expected Outcomes: The study is expected to demonstrate that Empower@Home, when supported by aging service providers, is more effective and cost-effective than enhanced usual care in reducing depressive symptoms and improving other psychosocial outcomes. Additionally, the findings will provide valuable insights into the barriers and facilitators to implementing DMHIs in community settings, offering guidance for future scalability and sustainability of such interventions.

Innovation: Empower@Home integrates user-centered design principles, community participatory research, and innovative engagement strategies, such as character-driven storytelling, to enhance user experience and therapeutic outcomes. The use of aging service providers as lay coaches not only addresses the shortage of mental health professionals but also aligns with the existing infrastructure of aging services, making the program highly scalable and sustainable.

This trial will contribute significantly to the growing body of evidence on the effectiveness of DMHIs in real-world settings and inform strategies for broader implementation within community-based aging services.

ELIGIBILITY:
Inclusion Criteria:

* (1) be receiving or eligible to receive services at the recruitment sites
* (2) read and speak English
* (3) be at least 50 years old
* (4) have at least moderate depressive symptoms at screening (≥ 8 on the Patient Health Questionnaire-9 [PHQ-9]).
* (5) Participants who are NOT currently receiving outside therapy must agree NOT to start outside therapy during study participation. Participants who are currently receiving outside therapy must agree NOT to increase their outside therapy frequency during study participation.

Exclusion Criteria:

* (1) probable dementia based on the Blessed Orientation and Memory Scale.
* (2) moderate or high risk of suicide based on the 6-item Columbia-Suicide Severity Rating Scale
* (3) a terminal illness with less than six months to live or unstable physical health conditions based on self-report
* (4) a diagnosis of a psychotic disorder like schizophrenia or bipolar disorder based on self-report and medical chart review
* (5) severe vision impairment based on self-report (i.e., legally blind)
* (6) current substance use disorders or receiving substance use treatment.
* (7) currently receiving outside therapy more frequently than once a month or have started a new therapy treatment less than 3 months ago

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 9 item standardized measures of depressive symptom severity. PHQ-9 score ranges from 0 to 27, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in Duke Social Support Index (DSSI)-10 | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 10 item standardized measure for social interaction and satisfaction with social support. Total score ranges from 10 to 30, higher score means higher social support.
Change in EuroQol 5-Dimension 5-level (EQ-5D-5L) | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 5 item standardized quality of life measure. EuroQol 5-Dimension 5-level is a commonly used tool to measure health-related quality of life. The final index score for the EQ-5D-5L is calculated by converting the health states described by a respondent into a single summary index value using a scoring algorithm. The EQ-5D-5L index score typically ranges from less than 0 (worse than death) to 1 (perfect health).
Change in Hamilton Depression Rating Scale (HAM-D) | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 7-item clinician-administered assessment of depression. HAM-D is a clinician-administered interview commonly used to assess depressive symptoms and will be administered by a Master of Social Work-prepared research staff who will complete the HAMD training offered by the Center for Telepsychology. Total scores range from 0 to 26, with a higher score indicating more severe symptoms.
Change in WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change from Baseline at 12, 24, and 36 weeks
  Change in 12 item standardized measure for health and disability. The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) is a standardized tool developed by the World Health Organization for measuring health and disability across different cultures and settings. It captures the impact of a health condition on daily life across six domains: cognition, mobility, self-care, getting along with people, life activities, and participation in society. Total scores range from 0 to 60, higher scores means greater level of disability or loss of function.
Change in Pain intensity assessed by the Pain, Enjoyment, and General Activity (PEG) Scale | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 3-item measure of chronic pain. The PEG Scale (Pain, Enjoyment, General Activity) is a brief, self-reported measure assessing three dimensions of chronic pain: pain intensity, the degree to which pain interferes with enjoyment of life, and the extent of its interference with general activity. Total scores range from 0 to 10, higher score means worse pain and more severe interference with life and activities.
Change in Generalized Anxiety Disorder Assessment-7 (GAD-7) | Change from Baseline to follow-up assessments at 12, 24, and 36 weeks
  Change in 7-item standardized measure for severity of anxiety symptoms. GAD-7 score ranges from 0 to 21, higher score means more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared through the National Institute of Mental Health's (NIMH) Data Archive (NDA), in compliance with NIMH funding requirements. The data will be available to qualified researchers following appropriate data use agreements. All quantitatively collected, non-identifying IPD, along with data dictionaries will be deposited to the NDA.
Supporting Information: ICF
Time Frame: Aligning with NIMH guidelines, all final IPD and supporting information will be deposited to NDA within one year of study completion.
Access Criteria: Researchers will apply for data access via the NDA.
URL: https://nda.nih.gov/nda/data-contribution

REFERENCES:
- [Derived] Xiang X, Narbut E, Zhang X, Ash S, Turner S, An R, Jester JM, Park S, Habash S, Himle JA. Leveraging Aging Service Providers to Support Internet-Based Cognitive Behavioral Therapy for Depression in Homebound Older Adults: Protocol for a Type 1 Hybrid Effectiveness-Implementation Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 5;14:e72953. doi: 10.2196/72953. PMID 40910699
- See also: Intervention website — https://empower-at-home.com/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT06584422/ICF_001.pdf